Official Title:

Cerebral Venous Thrombosis Cohort Study in China Mainland.

Document date:

4/16/2019

Statistical analysis plan:

Unpaired t-test was used to compare the continuous variables between two subgroups. Variance analysis was used to compare the continuous variables among three or more groups. If the dependent variable is a continuous variable, the influence of the independent variable on the dependent variable is analyzed by linear regression. If dependent variables are classified variables, the influence of independent variables on dependent variables is analyzed by binary or multivariate logistic regression. Chi-square test was used to compare frequency, percentage and incidence. P < 0.05 is defined as statistical significance.